CLINICAL TRIAL: NCT05843214
Title: Transcranial Doppler, Optic Nerve Envelope Diameter and Quantitative Pupillometry Measurements in Postoperative Resuscitation Neurosurgery
Brief Title: Transcranial Doppler, Optic Nerve Envelope Diameter and Quantitative Pupillometry Measurements
Acronym: DOPPLER
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Other Study IDs: 2021/CHU/04
Record Dates: First submitted 2023-04-11; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Neurological Complication
MeSH Terms: interventions — Ultrasonography, Doppler, Transcranial

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Non-invasive neuromonitoring evaluation (transcranial doppler, optic nerve envelope diameter and quantitative pupillometry) — 4 days Post-operation follow-up. Data will be gathered before the surgery and at regular times after the surgery until day 4

SUMMARY:
Non-invasive neuromonitoring tools such as transcranial doppler, optic nerve envelope diameter measurement and quantitative pupillometry are routinely used in acute brain injured patients as part of multimodal neuromonitoring with the aim, among others, of detecting episodes of intracranial hypertension, each method allowing the study of one of the different pathophysiological mechanisms of its impact.

However, at present there is no data in the literature on the value of these non-invasive neuromonitoring tools in the management of patients undergoing controlled intracranial surgery.

The study aims to help the early detection of postoperative neurological deterioration.

ELIGIBILITY:
Inclusion Criteria:

* Regulated intracranial surgery: scheduled > 48 hours
* French-speaking patient
* No opposition from the patient or a relative when the patient is unable to consent

Exclusion Criteria:

* Chronic subdural haematoma
* Isolated cerebral endovascular procedure
* Stereotactic biopsy
* Scheduled ventriculoperitoneal shunt or isolated ventriculocisternostomy
* Specific non-inclusion criteria for quantitative pupillometry: known pupillary abnormalities, glaucoma, cataract surgery and any ocular surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing planned neurosurgery
Sampling Method: Non-Probability Sample
Enrollment: 230 (Estimated)
Dates: Start 2023-02-10 (Actual); Primary Completion 2026-02-09 (Estimated); Study Completion 2026-06-09 (Estimated)

PRIMARY OUTCOMES:
Evolution of non-invasive neuromonitoring measures (using transcranial doppler) | From 1 hour before the surgery until Day 4 post-surgery
  This emasure will be performed bilaterally at the level of the first part of the middle cerebral artery, the values collected will be:
  * Systolic, mean and diastolic velocities; pulsatility index
  * Estimation of intracranial pressure
Evolution of non-invasive neuromonitoring measures (optic nerve envelope diameter) | From 1 hour before the surgery until Day 4 post-surgery
  The diameter of the optic nerve envelope will be collected bilaterally using an ultrasound machine
Evolution of non-invasive neuromonitoring measures (quantitative pupillometry) | From 1 hour before the surgery until Day 4 post-surgery
  The values collected will be :
  - Size, quantification of the amplitude of variation to light, latency and speed of constriction of the pupil, presence or absence of anisocoria (defined by a difference >1mm in size between the two pupils)

CONTACTS AND LOCATIONS:
Overall Officials: Romain ASMOLOV, MD, Principal Investigator — CHU de la Réunion
Locations (1):
- CHU de la Réunion, Saint-Pierre, Reunion

IPD SHARING:
Plan to Share IPD: No